CLINICAL TRIAL: NCT02261259
Title: Effects of Osteopathic Manipulative Treatment on Neuromuscular Control of the Head-neck System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jacek Cholewicki, Walter F. Patenge Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NCCAM U19 AT006057 Project 3; 5U19AT006057-02 (NIH)
Record Dates: First submitted 2014-09-19; First posted 2014-10-10 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate treatment (Experimental): This arm receives osteopathic manipulative treatment shortly after enrollment
  Interventions: Procedure: Osteopathic manipulative treatment
- Delayed treatment (Experimental): This arm receives osteopathic manipulative treatment approximately 4 weeks after enrollment
  Interventions: Procedure: Osteopathic manipulative treatment
- Healthy control (no neck pain) (No Intervention): In this arm, healthy controls are tested at baseline.

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment — Up to 4 sessions of osteopathic manipulative treatment (once per week)
  Arms: Delayed treatment; Immediate treatment

SUMMARY:
The overall goal of this project is to develop sensitive and objective clinical research tools for the assessment of head-neck motor control. In order to accomplish this goal, the investigators aim to quantify changes in head-neck motor control before and after osteopathic manipulative treatment. The investigators hypothesize that head-neck motor control will improve in neck pain participants after 4-weeks of treatment. Additionally, the investigators will compare position and force head-neck motor control between healthy controls and neck pain patients. The investigators hypothesize that baseline tests of position and force head-neck motor control will be better in healthy individuals than neck pain patients.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the inclusion criteria to participate in the study. Below is a list of inclusion criteria for ALL participants:

* Age 21-65 years
* Independently ambulatory
* Able to speak and read English
* Able to understand study procedures and to comply with them for the entire length of the study.

Below is an additional list of inclusion criteria for NECK PAIN participants:

* Willing to be randomized to either immediate or delayed treatment group.
* Musculoskeletal pain - primarily in the cervical region lasting longer than 3 months
* Pain rating greater than or equal to 3 out of 10 as indicated on the Numeric Rating Scale for Pain
* Neck Disability greater than or equal to 30% as indicated on the Neck Disability Index

Exclusion Criteria:

All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation. Exclusion criteria will be self-reported. However, during each treatment session, the physicians will be watching for clinical signs and symptoms not consistent with physical findings that are suggestive of the presence of any of the exclusion criteria. In such a case, further treatment will be discontinued and the subject will be excluded.

Below is a list of exclusion criteria for ALL participants:

* Inability or unwillingness of individual to give written informed consent.
* Physical therapy or any other form of manual medicine (e.g., Osteopathic Manipulative Medicine, Chiropractic Manipulation, etc.), acupuncture or spinal injections within one month prior to study enrollment
* Workers' compensation benefits in the past 3 months or ongoing medical legal issues
* Possibly pregnant
* Extreme obesity (BMI>36)
* Currently using electrical implants (e.g., cardiac pacemakers, drug delivery pumps, etc.)

History of:

* Spinal surgery
* Spinal fracture
* Spinal infection (e.g., osteomyelitis)
* Cancer

Unresolved symptoms from:

* Head trauma
* Inner ear infection with associated balance and coordination problems
* Orthostatic hypotension
* Uncontrolled hypertension
* Vestibular disorder (e.g. vertigo)

Current diagnosis of:

* Significant spinal deformity (e.g., scoliosis > 20 degrees, torticollis)
* Ankylosing spondylitis
* Spondylolisthesis grades III or IV
* Rheumatoid arthritis
* Osteoporosis
* Angina or congestive heart failure symptoms
* Active bleeding or infection in the back
* Blindness
* Seizures
* Neurologic disease (e.g., Parkinson's disease, multiple sclerosis, cerebral palsy, Alzheimer's disease, amyotrophic lateral sclerosis, stroke or transient ischemic attack in the past year, cervical dystonia)

Conditions recognized by a physician any time during the study:

* Significant or worsening signs of neurologic deficit
* Symptoms are not consistent with mechanical findings
* Other conditions impeding protocol implementation

Below is an additional exclusion criterion for healthy control participants:

• Based on the minimal clinically important difference of 2 points (Childs et al., 2005), "healthy controls" with 2 points or greater pain on NRS will not be eligible to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 4 and from week 4 to 8 in head position tracking accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be seated in an upright position with their upper body secured to a backrest and will wear a head harness with an attached position sensor. The angular position of the head will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by moving their head. Accuracy will be determined by taking the difference between the target position signal and the actual head position (measured in degrees with string potentiometers).
Change from baseline to week 4 and from week 4 to 8 in head force tracking accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be seated in an upright position with their upper body secured to a backrest and will be asked to generate force with their head against a fixed pad. The pad will be attached to a load cell that monitors how much force is being generated by their head. The force level will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by generating force with their head. Accuracy will be determined by taking the difference between target force signal and the actual head force (measured in Newtons with the load cell).
Change from baseline to week 4 and from week 4 to 8 in head position stabilization accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be sitting upright in a seat mounted to a robotic platform (Mikrolar Hexapod Robot) with their upper body secured to a backrest and will wear a head harness with an attached position sensor. The robotic platform will provide an angular perturbation to the participant about the cervical spine in the sagittal plane while the participant is asked to maintain (stabilize) their head position in the upright posture. Accuracy will be determined by measuring the amount of head displacement (measured in degrees with string potentiometers) during the perturbation trial.
Change from baseline to week 4 in neck force and muscle activation directionality | Change from baseline to week 4
  Participants will be seated in an upright position with their upper body secured to a backrest and will be asked to generate force with their head against a fixed pad. They will be asked to performed 6-seconds isometric exertions in different directions. Surface EMG will be recorded from the sternocliedomastoid, splenius capitis, and upper trapezius muscles. Muscle directionality will be determined by the EMG magnitude in each direction of exertion.
Change from week 4 to 8 in neck force and muscle activation directionality | Change from week 4 to 8
  Participants will be seated in an upright position with their upper body secured to a backrest and will be asked to generate force with their head against a fixed pad. They will be asked to performed 6-seconds isometric exertions in different directions. Surface EMG will be recorded from the sternocliedomastoid, splenius capitis, and upper trapezius muscles. Muscle directionality will be determined by the EMG magnitude in each direction of exertion.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in physical function, anxiety, depression, fatigue, sleep, satisfaction with social role, and pain with PROMIS-29 questionnaire.
Change in concomitant medication | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in the use of medication for treating neck pain, including the type of medication and the quantity of medication (i.e., number of pills) with a questionnaire.
Change in neck disability | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in functional activities related to neck disability with the Neck Disability Index questionnaire.
Change in fear avoidance behavior | The expected average is weekly for this outcome measure until the end (expected average of 8 weeks).
  Assesses weekly changes in fear avoidance behavior using the Fear Avoidance Beliefs questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Cholewicki, PhD, Principal Investigator — Michigan State University; Norman P Reeves, PhD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - MSU Osteopathic Manual Medicine, East Lansing, Michigan
  - MSU Musculoskeletal Rehabilitation, Lansing, Michigan
  - Michigan State University Center for Orthopedic Research, Lansing, Michigan

REFERENCES:
- [Background] Reeves NP, Popovich JM Jr, Priess MC, Cholewicki J, Choi J, Radcliffe CJ. Reliability of assessing trunk motor control using position and force tracking and stabilization tasks. J Biomech. 2014 Jan 3;47(1):44-9. doi: 10.1016/j.jbiomech.2013.10.018. Epub 2013 Oct 22. PMID 24262851
- See also: Website for Michigan State University Center for Orthopedic Research — http://orthopedicresearch.msu.edu/
- See also: Website for the National Center for Complementary and Alternative Medicine (Sponsor) — http://nccam.nih.gov/